CLINICAL TRIAL: NCT02030028
Title: Open Label Study to Evaluate Efficacy and Safety of Short-Term, Adjunctive Adrenocorticotropic Hormone (ACTH) Gel in Rheumatoid Arthritis
Brief Title: ACTH Gel Therapy in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana Ascherman (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Dana Ascherman, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19050342
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Results first posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; ACTH gel
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACTHAR Gel (Other): Open label Adrenocorticotropic Hormone (ACTH) Gel for 12 weeks, 80u (1mL), given subcutaneously twice each week.
  Interventions: Drug: ACTHAR gel

INTERVENTIONS:
Drug: ACTHAR gel — Subjects are given the ACTHAR gel subcutaneously twice per week for 12 weeks.
  Other Names: Adrenocorticotropic hormone

SUMMARY:
The purpose of this research study is to evaluate if the study drug, ACTH Gel helps decrease the disease symptoms in people with Rheumatoid Arthritis (RA) who are already taking medications prescribed by their physician and are still experiencing disease symptoms.

ACTH gel has been a Food and Drug Administration-approved treatment for Rheumatoid Arthritis since 1952, and in 2010 the FDA retained RA as a disease approved for ACTH gel use. Despite its FDA approval there is very limited data on its how well ACTH gel works in improving the symptoms of people with RA.

DETAILED DESCRIPTION:
This study is for people who are currently taking a biologic therapy for Rheumatoid Arthritis and who are still experiencing symptoms. Subjects are given the ACTH gel to take twice each week for 12 weeks as a supplement to current therapies. Subjects are required to visit the clinic for a baseline visit, at 2 weeks, 4 weeks, 8 weeks and 12 weeks. We will obtain a blood sample for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* 18 year of age and older
* RA diagnosis by American College of Rheumatology criteria
* Active disease (CDAI > 10)
* Have received at least are biologic agent for at least 6 months
* May or may not be receiving oral daily steroids (less than or equal to 20 mg/day) of prednisone equivalent
* No current active infections requiring antibiotics
* Patients must be on stable doses of RA therapies (e.g., methotrexate or other RA therapies for at least 4 weeks prior to baseline visit)

Exclusion Criteria:

* Less than 18 years of age
* Unable or unwilling to give Informed Consent
* Have an active infection requiring the use of antibiotics
* Women who are pregnant
* Uncontrolled hypertension
* Abnormal renal function
* Abnormal liver function as defined by and increased Alanine transaminase (ALT,) and aspartate aminotransferase (AST) that is greater than 5 times normal.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry W Moreland, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No patients were excluded from the study based on enrollment criteria. Because ACTHAR administration was add on therapy, no wash out period was required.
Period: Overall Study
Arm/Group | ACTHAR Gel
Started | 18
Completed | 13
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — lack of transportation | 1

BASELINE CHARACTERISTICS:
Arm/Group | ACTHAR Gel
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 55.3 [35.7 to 68.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18
Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: mm/hr] — scale: 0 - >120 mm/hr (normal range 0-20)
  mm/hr | 37.2 (33.8)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/dl] — scale: continuous measure of serum C-Reactive Protein concentration from 0 mg/dl, with undefined upper limit (normal range 0-0.8 mg/dl)
  mg/dl | 0.42 (0.33)
Tender Joints [Median (Inter-Quartile Range); unit: joints] — scale: 0-28 joints
  joints | 6 [3.25 to 11.75]
Swollen Joints [Median (Inter-Quartile Range); unit: joints] — scale: 0-28 joints
  joints | 6 [5.25 to 9.75]
Physician Global Assessment of Disease Activity [Median (Inter-Quartile Range); unit: units on a scale] — scale: 0-10 cm (0=no disease activity, 10=maximal disease activity)
  units on a scale | 5 [4.125 to 5.5]
Patient Global Assessment of Disease Activity [Median (Inter-Quartile Range); unit: units on a scale] — scale: 0-10 cm (0=no disease activity, 10=maximal disease activity)
  units on a scale | 7 [6 to 9]
CDAI (Clinical Disease Activity Index) [Median (Inter-Quartile Range); unit: units on a scale] — scale: 0-76 based on composite of tender joint count (0-28), swollen joint count (0-28), patient global disease activity (0-10 cm), and physician global disease activity (0-10 cm). Higher numbers indicate greater/more severe disease activity.
  units on a scale | 27 [25.5 to 32.5]
DAS28-ESR (Disease Activity Score 28--ESR) [Mean (Standard Deviation); unit: units on a scale] — scale: based on composite of tender joints (0-28), swollen joints (0-28), patient assessment of disease activity (0-100 mm), and ESR (0 - >120)
  calculation of total score based on formula: 0.56*√(TJC28)+0.28*√(SJC28)+0.014*GH+0.70*ln(ESR)
  Total score range: 0 (minimum) to 9.2 (maximum); remission: < 2.6 low disease activity: 2.6-3.1 moderate disease activity: 3.1-5.1 high disease activity: >5.1
  units on a scale | 5.6 (1.6)
DAS28-CRP (Disease Activity Score 28--CRP) [Mean (Standard Deviation); unit: units on a scale] — scale: based on composite of tender joints (0-28), swollen joints (0-28), patient assessment of disease activity (0-100 mm), and CRP (0 - 150)
  calculation of total score based on formula: (0.56 × √TJC) + (0.28 × √SJC) + (0.014 × PGA [mm]) + (0.36 × ln(CRP in mg/L+1) + 0.96
  Range of total score: 0 (minimum) to 8.61 (maximum); remission: < 2.5 low disease activity: 2.5-2.9 moderate disease activity: 2.9-4.6 high disease activity: >4.6
  units on a scale | 4.2 (0.6)
fatigue severity scale--functional well-being subscale [Median (Inter-Quartile Range); unit: units on a scale] — scale: 0-28 based on 0 (not fatigued)-4 (very fatigued) Likert scale within 7 domains/questions; 0=limited fatigue, 28=high level of fatigue
  units on a scale | 13 [8.5 to 16.75]
FACIT (Functional Assessment of Chronic Illness Therapy) Fatigue Scale [Median (Inter-Quartile Range); unit: units on a scale] — Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale: 0-52 based on 0 (not fatigued)-4 (very fatigued) Likert scale within 13 domains/questions; 0=limited fatigue, 52=high level of fatigue
  units on a scale | 26 [18.5 to 34]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Clinical Disease Activity Index (CDAI) Between Week 0 and Week 12
Description: percentage of participants achieving >20% improvement in CDAI after 12 weeks of therapy (>20% reduction in CDAI relative to baseline based on ratio of CDAI at week 12 to CDAI at week 0: CDAI Week 12/CDAI Week 0 < 0.8 meets criteria for improvement, as lower CDAI scores represent lower disease activity)
Time Frame: 12 weeks
Population: Study completers (9/13 had evaluable data at baseline and week 12)
Measure: Count of Participants; unit: Participants
Arm/Group | ACTHAR Gel
Number analyzed (Participants) | 9
Participants | 8

2. Secondary Outcome: Change in the Disease Activity Score (DAS28-CRP) Between Week 0 and Week 12
Description: Change in the Disease Activity Score 28-CRP (DAS28-CRP) at week 12 relative to baseline (week 0), where lower DAS28-CRP scores at week 12 represent improvement.
  Scale: 0-8.61 (lower scores indicate reduced disease activity)
Time Frame: 12 weeks
Population: Study completers--5/13 with evaluable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ACTHAR Gel
Number analyzed (Participants) | 5
units on a scale | -0.87 (1.75)

3. Secondary Outcome: Changes in Acute Phase Reactants (CRP) Between Week 0 and Week 12
Description: Changes in C-reactive protein value (mg/dl): reduction in CRP values at week 12 relative to week 0 represents improvement (week 12 CRP-baseline CRP < 0))
Time Frame: 12 weeks
Population: Study completers--7/13 with evaluable data
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | ACTHAR Gel
Number analyzed (Participants) | 7
mg/dl | 0.36 (1.33)

4. Secondary Outcome: Change in Acute Phase Reactants (ESR) Between Week 0 and Week 12
Description: Change in ESR--reduction in ESR at week 12 relative to baseline (week 0) represents improvement (week 12 ESR - baseline ERS < 0)
Time Frame: 12 weeks
Population: Study completers--8/13 with evaluable data
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | ACTHAR Gel
Number analyzed (Participants) | 8
mm/hr | -7.38 (28.30)

5. Secondary Outcome: Patient Reported Changes in Fatigue Between Week 0 and Week 12
Description: The FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue) scoring metric assesses fatigue using 13 questions rated on a Likert scale of 0 (no fatigue)-4 (severe fatigue); total scores range from 0-52, with higher total scores representing more severe fatigue. The difference in FACIT-F scores between weeks 12 and week 0 (calculated as FACIT-F score week 12 minus FACIT-F score at week 0) indicates changes in fatigue relative to baseline, where reduction of FACIT-F score at week 12 represents improvement in fatigue.
Time Frame: 12 weeks
Population: Study completers--13/13 with evaluable data
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | ACTHAR Gel
Number analyzed (Participants) | 13
units on a scale | -3.8 [-23.1 to 5.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 16 week period spanning from baseline to 16 weeks
Description: No deviation from standard adverse events definitions
Arm/Group | ACTHAR Gel
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTHAR Gel (N=18)
rib fractures (Musculoskeletal and connective tissue disorders) | 1 (1) — ATV accident resulting in multiple rib fractures

LIMITATIONS AND CAVEATS:
This trial was limited by small sample size and reduced number of participants completing the study. Statistical analysis was compromised by missing standard-of-care laboratory values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT02030028/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT02030028/ICF_001.pdf